CLINICAL TRIAL: NCT05431881
Title: The Effect of Preoperative Binaural Sound on Propofol Dose Required for Induction of General Anesthesia: a Randomized, Placebo-controlled Trial
Brief Title: Binaural Sound Effects for General Anesthesia
Acronym: BS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jeong-Hwa Seo, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2204-007-1313
Record Dates: First submitted 2022-06-09; First posted 2022-06-24 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Anesthesia, General
Keywords: Propofol; Brain Waves

STUDY DESIGN:
Intervention Model Description: A prospective randomized study
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): A silent state (a wave file made without sound) is applied for at least 20 minutes from 20 minutes before arrival to the operating room. The sound generator is a smartphone device, set the volume (at a volume corresponding to 60 dB in the experimental group), and hang it on the transport bed. Upon arrival in the operating room, before anesthesia, the volume is adjusted to 0.
  Interventions: Procedure: Silent
- Binaural beat (Experimental): In the experimental group, the binaural sound, which was produced by the beat of 2Hz difference, is applied for 20 minutes from 20 minutes before arrival to the operating room. The sound generator is a smartphone device, set the volume corresponding to 60 dB, and hang it on the transport bed. Upon arrival in the operating room, before anesthesia, the volume is adjusted to 0.
  Interventions: Procedure: Binaural beat

INTERVENTIONS:
Procedure: Binaural beat — Different frequencies are transmitted in both ears, causing beats. The low frequency sound generated by beats induces brainwaves entrainment.
  Arms: Binaural beat
Procedure: Silent — Apply a wave file which is created in silence.
  Arms: Control

SUMMARY:
30 minutes before entering the operating room, the anxiety score is evaluated using a visual analogue scale (VAS) score, and stereo headphones, which can transmit binaural beat, are put on. According to a computer-generated assignment table, subjects are divided into an experimental group and a control group.

Binaural beat is applied to the experimental group for 20 minutes, and a silent state is applied to the control group for 20 minutes. After entering the operating room, electrocardiogram, pulse oxymetry, non-invasive blood pressure monitor, and sensor for depth of anesthsia are attached. Before induction of anesthesia, the anxiety score is evaluated on a VAS, again.

For anesthesia induction, propofol is administered at a rate of 10 mg every 15 seconds over 5 seconds. Assess the amount of propofol administered until the response to voice ("Open your eyes.") is absent, the subject's eyelash reflex disappears, and the PSI reaches below 50. Discontinue propofol injection when all three assessments (unresponsiveness to voice, loss of eyelash reflexes, Patient Sate Index (PSI) ≤ 50) become positive.

DETAILED DESCRIPTION:
30 minutes before entering the operating room, anxiety is evaluated on a VAS score (0-100mm, a ruler without scale) and stereo headphones, which can transmit binaural beat, are put on. A third party unrelated to the experiment sees the randomization table and applies binaural sound to the experimental group and silent state (silent sound file) to the control group for 20 minutes.

The sound generator is a smartphone device, which is hung on the transport bed. The volume is set to a level corresponding to 60dB.

After entering the operating room, start monitoring vital signs and depth of anesthesia (PSI) by attaching an electrocardiogram, pulse oxymetry, non-invasive blood pressure monitor, and sedline. Prepare by connecting a 3-way at the most proximal part of the intravenous cannula. After changing the volume to 0, take off the headphones, and evaluate the anxiety score using VAS.

Preoxygenation with oxygen 8L/min is sufficient, and in order to reduce venous pain caused by propofol injection, 1% lidocaine 50mg is pre-administrated. For anesthesia induction, 10mg propofol is administered every 15 seconds for 5 seconds. Assess the amount and time of propofol administered until the response to the voice ("Open your eyes.") is absent, the patient's eyelash reflex disappears, and the PSI reaches below 50. Propofol is administered until all three evaluations (no response to voice, loss of eyelash reflexes, PSI ≤ 50) are positive. After that, propofol is not administered. During anesthesia induction, the concentration of the inhaled anesthetic is adjusted so that Psi is between 25-50, and the anesthesia process is the same for both groups.

Continuously monitor blood pressure, pulse, and Psi, and record the MAC value of the inhaled anesthetic immediately after tracheal intubation, vital signs, and Psi.

The raw data of EEG is stored through the Sedline sensor and additionally analyzed and evaluated. The primary endpoint is the dose of propofol administered until the response to the voice ("Open your eyes.") is absent

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 20-50 who require general anesthesia
* Patients who are able to provide written consent to participate in the clinical trial, to understand the procedure of this clinical trial, and to fill out the questionnaire appropriately
* Patients with ASA physical status classification 1-2
* Patients weighing from 50 kg to 80 kg

Exclusion Criteria:

* Patients with hearing loss or using hearing aids
* Patients who received narcotic analgesics or sedative drugs within 1 week
* Patients with alcohol or drug dependence
* Patients with drug hypersensitivity to propofol
* Patients with arrhythmia, cardiovascular disease, and decreased heart function
* Patients with liver failure
* Patients who are judged to be inappropriate for this clinical trial according to the opinions of investigators

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-09-07 (Estimated); Study Completion 2023-10-07 (Estimated)

PRIMARY OUTCOMES:
Propofol dose | Until the response to the voice ("Open your eyes.") becomes absent (up to 5minutes)
  The amount of propofol administered until the response to the voice ("Open your eyes.") becomes absent

SECONDARY OUTCOMES:
Propofol dose | until eyelash reflex disappears (up to 5minutes)
  Propofol dose administered until eyelash reflex disappears
Propofol dose | until PSI falls below 50 (up to 5minutes)
  Propofol dose administered until PSI falls below 50
Anxiety | 20minutes before the entrance to the operating room
  Anxiety is evaluated using VAS score(0-100mm ruler without a scale), 20minutes before the entrance to the operating room
Anxiety | just before induction of anesthesia
  Anxiety is evaluated using VAS score(0-100mm ruler without a scale), just before induction of anesthesia
Brainwaves | From the time you enter the operation room until the anesthesia induction is complete (up to 30minutes)
  brainwaves (raw data) which are collected in the Sedline device

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Hwa Seo, MD.,PhD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Background] Schmid W, Marhofer P, Opfermann P, Zadrazil M, Kimberger O, Triffterer L, Marhofer D, Klug W. Brainwave entrainment to minimise sedative drug doses in paediatric surgery: a randomised controlled trial. Br J Anaesth. 2020 Sep;125(3):330-335. doi: 10.1016/j.bja.2020.05.050. Epub 2020 Jul 8. PMID 32653082
- [Background] Turkistani A, Abdullah KM, Al-Shaer AA, Mazen KF, Alkatheri K. Melatonin premedication and the induction dose of propofol. Eur J Anaesthesiol. 2007 May;24(5):399-402. doi: 10.1017/S0265021506001505. Epub 2006 Nov 10. PMID 17094871
- [Background] Facco E, Stellini E, Bacci C, Manani G, Pavan C, Cavallin F, Zanette G. Validation of visual analogue scale for anxiety (VAS-A) in preanesthesia evaluation. Minerva Anestesiol. 2013 Dec;79(12):1389-95. Epub 2013 Jul 9. PMID 23860442
- [Background] Padmanabhan R, Hildreth AJ, Laws D. A prospective, randomised, controlled study examining binaural beat audio and pre-operative anxiety in patients undergoing general anaesthesia for day case surgery. Anaesthesia. 2005 Sep;60(9):874-7. doi: 10.1111/j.1365-2044.2005.04287.x. PMID 16115248
- [Derived] Kim YJ, Choe HW, Yoon SB, Lee H, Kim HS, Seo JH. Effects of preoperative binaural beats on the propofol dose for induction of general anesthesia: a randomized controlled trial. Can J Anaesth. 2025 Jul;72(7):1101-1109. doi: 10.1007/s12630-025-02993-5. Epub 2025 Jun 25. PMID 40563070